CLINICAL TRIAL: NCT03690037
Title: Single Centre Randomised Controlled Trial to Assess the Effect of the Addition of Twenty-four Hours of Oral Tranexamic Acid Post-operatively to a Single Intra-operative Intravenous Dose of Tranexamic Acid on Calculated Blood Loss Following Primary Hip and Knee Arthroplasty.
Brief Title: Investigating the Effect of Intravenous and Oral Tranexamic Acid on Blood Loss After Primary Hip and Knee Arthroplasty
Acronym: TRAC-24
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15039DB - SW
Record Dates: First submitted 2017-12-05; First posted 2018-10-01 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Primary Total Knee Arthroplasty; Primary Total Hip Arthroplasty
Keywords: Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: A Phase IV, single centred, open label, parallel group, randomised controlled trial
Masking Description: Not Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Experimental): Intervention Group 1: 1g intravenous Tranexamic Acid 100 milligrams (MG)/ML peri-operatively plus 1g oral Tranexamic Acid 500mg Tablets every 8hrs for up to 24hrs
  Interventions: Drug: Tranexamic Acid 100 MG/ML; Drug: Tranexamic Acid 500 MG
- Intervention Group 2 (Experimental): Intervention Group 2: 1g intravenous Tranexamic Acid 100 MG/ML peri-operatively
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- Control Group 3 (No Intervention): Standard care - no TXA

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — Tranexamic Acid: 100 MG/ML Solution for injection
  Other Names: TXA
  Arms: Intervention Group 1; Intervention Group 2
Drug: Tranexamic Acid 500 MG — Tranexamic Acid: Tranexamic Acid 500mg Tablets
  Other Names: TXA
  Arms: Intervention Group 1

SUMMARY:
Patients having a hip or knee replacement can lose almost a third of their blood during and after the operation. Many patients, especially those who are older will need a blood transfusion, suffer from anaemia, or have a slow recovery after the operation. Tranexamic acid is a medication used to treat or prevent excessive blood loss, but in joint replacements, is only used in patients who are likely to bleed a lot. This trial aims to find out how well tranexamic acid works to reduce blood loss after the operation in a large group of patients having a hip or knee replacement, including those at risk of blood clots. This study also aims to find out how safe tranexamic acid treatment is to use in different patients and the best way to give tranexamic acid (in tablet form or through a drip), as well as how much to give and how long it should be given after an operation. All adults awaiting non-emergency hip or knee replacement surgery will be considered.

Patients who are suitable and agree to take part are randomly placed in one of two treatment groups: receiving tranexamic acid during the hip or knee operation through a drip, or receiving treatment during the hip or knee operation through a drip plus taking a tablet every 8 hours up to 24 hours after the operation. Initially, a no treatment group was included, however, one year after the trial started, the Data Monitoring and Ethics Committee who check safety, advised to stop allocation of patients to the no treatment group.

For all patients, blood loss is recorded up to 48 hours after surgery. Blood samples are also taken in order to measure how well the heart and blood clotting systems are working. If the routine kidney function tests taken before the operation show less than normal function, a lower dose of tranexamic acid is used.

It is expected that patients who receive the tranexamic acid will lose much less blood during and after their operation, and so be less likely to need a blood transfusion, have reduced stress on the heart and have an easier recovery. It is thought that patients with a history of clots are more likely to have another clot when taking tranexamic acid. Therefore, this trial will include these patients to try and find out if this is true as these patients will benefit the most from reduced blood loss.

DETAILED DESCRIPTION:
Although numerous studies have demonstrated efficacy in using tranexamic acid (TXA) in primary hip and knee arthroplasty, it has not yet become a recognised standard of care in the United Kingdom (UK). In part, this is because trials to date have excluded many of the patients who could most benefit from a reduced peri-operative blood loss. This trial aims to maximize the potential of TXA by continuing administration post-operatively, at the time of greatest loss. In doing so, the aim is to establish a standardised protocol that can be adopted by other units. Also, despite any published evidence and the excellent safety profile of TXA, there have been concerns about a potential increased risk of venous thrombo-embolism (VTE) which in itself has been a contentious issue in the UK. The exclusion criteria have been adapted in this trial to address these safety concerns.This trial will contribute to establishing the effect of TXA on perioperative blood loss.

Reducing blood loss after hip and knee arthroplasty helps patients avoid anaemia and allogenic blood transfusion with their incumbent risks. TXA is effective intravenously and topically at reducing perioperative bleeding in various surgeries, the evidence in joint arthroplasty is compelling with calculated blood losses reduced by 30% and the need for a transfusion by 50%. However, it remains unclear as to whether extending a dosing regime of TXA beyond the immediate perioperative period would lead to further reductions in blood loss. Oral TXA would be a cheaper and less labour intensive mode of delivery post-operatively than either intravenous bolus or intravenous infusion regimes.

Patients undergoing joint arthroplasty are often elderly with co-morbidities; this frailty makes them particularly vulnerable to the adverse effects of major blood loss. Reducing bleeding in this group is likely to be particularly beneficial to patient outcomes.The majority of blood loss occurs in the first 24 hours post-operatively. A dosing regimen of intravenous TXA eight hourly for twenty-four hours has been suggested. Replacing this with an oral dose would be cheaper, less labour intensive for nursing staff and less disruptive for patients. One gram of oral TXA given 8 hourly for four doses following arthroplasty is consistent with prescribing guidance in the Summary of Product Characteristics (SPC) for local fibrinolysis.There is no evidence in the context of joint replacements to favour either 8 hourly or 6 hourly dosing. Both are licensed regimens as per SPC and therefore an 8 hourly regime is considered less intrusive to the patient.

Intravenous (IV) TXA has an elimination half-life of 3 hours (almost completely excreted unchanged in urine). Five hours after a dose of 10mg/kg IV bolus, the serum level is 5µg/L and it is thought that a level of 10µg/L provides 80% inhibition of fibrinolysis and is considered clinically effective. Oral TXA has a peak level 2 hours following ingestion. By administering the dose in the recovery ward 2 hours following knife to skin (KTS), this will give its peak effect just over 4 hours after the IV dose is administered in both hip and knee arthroplasty.

The aim is to minimise sub therapeutic TXA levels at the time of the highest bleeding risk. Nilsson (1987) noted that after total hip arthroplasty (THA), blood loss from drains was lower following a single 10mg/kg bolus intra-operatively in the first 2 hours but that the drain outputs then equilibrated between the TXA group and the control group after that for the following 10 hours. This supports the current hypothesis that administering further doses of TXA early post-operatively could further reduce blood loss. Also it will be easier to ensure accurate time of the first dose administration in recovery rather than on the ward due to greater staff availability.

This study initially used two tranexamic acid intervention groups (Groups 1 & 2) and one no treatment comparator group (Control Group 3). Although the benefits of using TXA in elective hip and knee arthroplasty to reduce blood loss has been shown, it has not become standard of care in the UK and hence the initial need for the Control Group 3. Following an interim analysis, it was recommended to stop randomisation to Control Group 3.

In addition, this study will incrementally contribute to the growing data relating to use of TXA in patients with a history of VTE. However, to definitively determine what impact TXA has on VTE in the peri-operative period would require a large appropriately powered multi-centre study.

Study Aim and Objectives

This is a Phase IV, single centred, open label, parallel group, randomised controlled trial involving primary hip and knee arthroplasty patients.

The overall aim of this study is to reduce blood loss in THA and Total Knee Arthroplasty (TKA) patients using TXA. While TXA has been shown to reduce blood loss in THA/TKA patients, the optimum method of delivery, optimum number of doses and optimum period of use is not clear. A previous audit of patients under the care of the Chief Investigator demonstrated that 5/6 of the blood loss occurs post wound closure. Therefore, hypothetically if TXA is given to a patient for over 24 hours following surgery it should further reduce blood loss as compared to TXA dosing in the immediate peri-operative period.

-Primary Objective: The primary objective is to determine if the use of oral TXA post-operatively for up to 24 hours will confer a reduction in the calculated blood loss at 48 hours beyond an intra-operative intravenous bolus alone for patients undergoing unilateral primary total hip or knee replacement.

-Secondary Objective: The secondary objective is to determine if the addition of oral TXA post-operatively to an intra-operative intravenous bolus of TXA produces any change in other measurable parameters as compared to those observed either with an intra-operative intravenous bolus alone or no TXA for patients undergoing unilateral primary THA/TKA.

While this study is not powered to answer questions such as whether the use of TXA can lower complications, it is important that complications are reported on. If it was found that using TXA increased the number of complications, this would be a clinically important outcome which should be reported.

Eligible participants were initially allocated to Intervention Group 1 (IV TXA peri-operatively plus 1g oral TXA every 8hrs for up to 24hrs), Intervention Group 2 (IV TXA peri-operatively) or Control Group 3 (standard care) with an allocation ratio of 2:2:1.

Patients with a renal impairment receive a reduced dose dependent on pre-operative serum creatinine.

Following the interim analysis it was recommended to stop randomisation to Control Group 3. Eligible participants are allocated to Intervention Group 1 or Intervention Group 2 with an allocation ratio of 1:1.

Anaesthetists, surgeons, other theatre, recovery and ward staff will not be blinded to the treatment, nor will the study investigators or the patient themselves.

However, the number of patients falling below the transfusion trigger will be blinded.The transfusion trigger will be set as per standardised protocol after consent and prior to randomisation. Therefore, the decision about whether or not to transfuse will not be blinded but the transfusion trigger will be blinded.

Staff in an off-site laboratory who are processing the blood samples will be blinded to the treatment Group allocation.

The TRAC-24 trial initially required a minimum of 1166 patients to be recruited. Recruitment was due to stop when 583 participants had been recruited for both the TKA and THA patients. However, following the interim analysis, randomisation of patients to Control Group 3 was stopped. Recruitment will now continue until a minimum of 932 patients, comprising of 466 TKA and 466 THA, is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Awaiting primary elective hip or knee replacement
2. ≥ 18 years of age and ≤100 years

Exclusion Criteria:

1. Patients who do not pass a pre-operative assessment for elective total hip or knee arthroplasty (THA/TKA)
2. Fractured neck of femur
3. Haemophiliac or coagulation disorders that require TXA
4. Allergy to tranexamic acid or any of its excipients
5. Platelets less than 75,000/mm3 at pre-operative assessment*
6. Patients on active treatment for venous thromboembolism (VTE) (deep vein thrombosis (DVT), pulmonary embolisms (PE)) within 6 months of surgery*
7. History of VTE within 6 months of surgery*
8. Patients who have had a myocardial infarction (MI) within 12 months*
9. Cardiac stent within 12 months of surgery*
10. Patients who have had a stroke (cerebrovascular accident (CVA)) or transient ischemic attack (TIA) within 9 months of surgery*
11. Use of antiplatelet medication within 7 days of surgery* (Does not include aspirin if dose <300mg).
12. Direct thrombin inhibitors within 2 days of surgery*
13. Factor Xa inhibitors within 2 days of surgery*
14. The International normalized ratio (INR) level is greater than or equal to 1.5 in a patient who has stopped warfarin in preparation for surgery
15. Hepatic failure*
16. Patients with epilepsy
17. Patients requiring therapeutic anticoagulation post-operatively e.g. Metallic heart valves.
18. Pregnant women, women who have not yet reached the menopause (no menses for ≥ 12 months without an alternative medical cause) who test positive for pregnancy or are unwilling to take a pregnancy test prior to trial entry
19. Patients who have been using Combined hormonal contraception (which includes combined oral contraception (COC), combined contraceptive transdermal patch and vaginal ring) within 4 weeks of surgery*.
20. Female patients who are breastfeeding
21. Treated with any other investigational medication or device within 60 days
22. Patients unable to provide informed consent
23. Patients who are unable or unwilling to commit to the study schedule of events
24. Patients unwilling to provide informed consent
25. Patients who present for simultaneous bilateral THA or TKA
26. Patients who are on renal dialysis and have an arteriovenous (AV) fistula
27. Patients who previously have been enrolled in this study

    * These are patients with contra-indications to primary hip or knee replacement.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Total Indirect blood loss | At 48 hours
  Volume (ml) of the total indirect blood loss at 48 hours

SECONDARY OUTCOMES:
Incidence of Post-operative haemoglobin falling below the transfusion trigger | Prior to discharge, up to 48 hours
  Incidence of post-operative haemoglobin falling below the transfusion trigger
Effect of body mass index (BMI) on the volume of indirect blood loss | At 48 hours post-surgery
  Effect of BMI on volume of indirect blood loss at 48 hours post surgery
Change in c-reactive protein | Pre-surgery to 48 hours post-surgery
  Change in c-reactive protein from pre-surgery to 48 hours post surgery
Change in Creatinine level | pre-surgery to 48 hours post-surgery
  Change in creatinine level from pre-surgery to 48 hours post surgery
Mortality | 90 days and 1 year post surgery
  Incidence of mortality at 90 days and 1 year

OTHER OUTCOMES:
Comparison of intra-operative blood loss between the groups | At 48 hours post surgery
  Comparison of intra-operative blood loss between the groups at 48 hours
Number of wound dressing changes in the 48 hours post surgery | 48 hours post-surgery
  Number of wound dressing changes
The number of requests for Post-operative Troponin levels prior to discharge | Tested prior to discharge up to Day 4 post-operative
  Number of requests (and the result) for post-operative troponin levels
Length of hospital stay after surgery | Up to 30 days
  Length of hospital stay after surgery in days
Incidence of allogenic blood transfusion prior to discharge from hospital | Tested prior to discharge up to Day 4 post-operative
  Incidence of allogenic blood transfusion prior to discharge from hospital
Incidence of allogenic blood transfusion within 90 days of surgery | 90 days post-surgery
  Incidence of allogenic blood transfusion within 90 days of surgery
Incidence of post-operative haemoglobin falling below transfusion trigger without patient being transfused up until time of discharge | Up to Day 4 post-operative
  Incidence of post-operative haemoglobin falling below transfusion trigger without patient being transfused
Incidence of post-operative arrhythmia within 90 days of surgery | within 90 days of surgery
  Incidence of post-operative arrhythmia within 90 days of surgery
Incidence of Pulmonary Embolism (PE) within 90 days of surgery | within 90 days of surgery
  Incidence of Pulmonary Embolism (PE) within 90 days of surgery
Incidence of proximal Deep Vein Thrombosis (DVT) within 90 days of surgery | within 90 days of surgery
  Incidence of proximal Deep Vein Thrombosis (DVT) within 90 days of surgery
Incidence of myocardial infarction within 90 days of surgery | 90 days post-surgery
  Incidence of myocardial infarction within 90 days of surgery
Incidence of stroke within 90 days of surgery | 90 days post-surgery
  Incidence of stroke within 90 days of surgery
Number of emergency hospital admissions or unplanned critical care admissions within 90 days of surgery | 90 days post-surgery
  Number of emergency hospital admissions or unplanned critical care admissions within 90 days of surgery
Number of returns to theatre for wound problems within 90 days of surgery | 90 days post-surgery
  Number of returns to theatre for wound problems within 90 days of surgery
Difference in indirect blood loss at 48 hours between patients on aspirin as a VTE prophylaxis compared with those on clexane | at 48 hours
  Difference in indirect blood loss at 48 hours between patients on aspirin as a VTE prophylaxis compared with those on clexane
Difference in indirect blood loss at 48 hours between patients placed in flexion in a knee jig for 6 hours post-operatively as opposed to those placed in flexion on a pillow | at 48 hours
  Difference in indirect blood loss at 48 hours between patients placed in flexion in a knee jig for 6 hours post-operatively as opposed to those placed in flexion on a pillow
Difference in indirect blood loss at 48 hours between patients in whom a tourniquet was used as compared to those in whom a tourniquet was not used during TKA | at 48 hours
  Difference in indirect blood loss at 48 hours between patients in whom a tourniquet was used as compared to those in whom a tourniquet was not used during TKA
Change on Oxford Hip Score (OHS) or Oxford Knee Score (OKS) from pre surgery to 90 days post-surgery | from pre surgery to 90 days post-surgery
  Change in total score in Oxford Hip Score or Oxford Knee Score which assess function and pain in patients undergoing hip or knee surgery
Change on Oxford Hip Score (OHS) or Oxford Knee Score (OKS) from pre surgery to 1 year post-surgery | from pre-surgery to 1 year post-surgery
  Change in total score in Oxford Hip Score or Oxford Knee Score which assess function and pain in patients undergoing hip or knee surgery
Differences in hospital costs associated with each treatment group | Up to 90 days
  Difference in cost associated with hospital stay between groups

CONTACTS AND LOCATIONS:
Overall Officials: David Beverland, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Primary Joint Unit, Musgrave Park Hospital, BHSCT, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Requests for data sharing will be reviewed on an individual basis by the Chief Investigator (CI) and Trial Management Group (TMG).

REFERENCES:
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] OKAMOTO S, SATO S, TAKADA Y, OKAMOTO U. AN ACTIVE STEREO-ISOMER (TRANS-FORM) OF AMCHA AND ITS ANTIFIBRINOLYTIC (ANTIPLASMINIC) ACTION IN VITRO AND IN VIVO. Keio J Med. 1964 Dec;13:177-85. doi: 10.2302/kjm.13.177. No abstract available. PMID 14279228
- [Background] Melander B, Gliniecki G, Granstrand B, Hanshoff G. Biochemistry and toxicology of amikapron; the antifibrinolytically active isomer of AMCHA. (A comparative study with epsilon-aminocaproic acid). Acta Pharmacol Toxicol (Copenh). 1965;22(4):340-52. doi: 10.1111/j.1600-0773.1965.tb01829.x. No abstract available. PMID 5898250
- [Background] Nilsson L, Rybo G. Treatment of menorrhagia with epsilon aminocaproic acid. A double blind investigation. Acta Obstet Gynecol Scand. 1965;44(3):467-73. doi: 10.3109/00016346509155880. No abstract available. PMID 5324474
- [Background] Shakur H, Elbourne D, Gulmezoglu M, Alfirevic Z, Ronsmans C, Allen E, Roberts I. The WOMAN Trial (World Maternal Antifibrinolytic Trial): tranexamic acid for the treatment of postpartum haemorrhage: an international randomised, double blind placebo controlled trial. Trials. 2010 Apr 16;11:40. doi: 10.1186/1745-6215-11-40. PMID 20398351
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Mitra B, Mazur S, Cameron PA, Bernard S, Burns B, Smith A, Rashford S, Fitzgerald M, Smith K, Gruen RL; PATCH-Trauma Study Investigators. Tranexamic acid for trauma: filling the 'GAP' in evidence. Emerg Med Australas. 2014 Apr;26(2):194-7. doi: 10.1111/1742-6723.12172. PMID 24708011
- [Background] Wishart N, Beaumont R, Young E, Mccormack V, Swanson M. 11th Annual Report- National Joint Registry. 2014;(December 2013).
- [Background] Frisch NB, Wessell NM, Charters MA, Yu S, Jeffries JJ, Silverton CD. Predictors and complications of blood transfusion in total hip and knee arthroplasty. J Arthroplasty. 2014 Sep;29(9 Suppl):189-92. doi: 10.1016/j.arth.2014.03.048. Epub 2014 May 24. PMID 25007727
- [Background] Krebs V, Hozack WJ, Callaghan JJ, Bohannon Mason J, Mont M, Parvizi J. Eliminating transfusion in primary joint arthroplasty-an achievable goal. J Arthroplasty. 2014 Aug;29(8):1511. doi: 10.1016/j.arth.2014.07.014. No abstract available. PMID 25085212
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Tan J, Chen H, Liu Q, Chen C, Huang W. A meta-analysis of the effectiveness and safety of using tranexamic acid in primary unilateral total knee arthroplasty. J Surg Res. 2013 Oct;184(2):880-7. doi: 10.1016/j.jss.2013.03.099. Epub 2013 Apr 25. PMID 23643299
- [Background] Molloy DO, Archbold HA, Ogonda L, McConway J, Wilson RK, Beverland DE. Comparison of topical fibrin spray and tranexamic acid on blood loss after total knee replacement: a prospective, randomised controlled trial. J Bone Joint Surg Br. 2007 Mar;89(3):306-9. doi: 10.1302/0301-620X.89B3.17565. PMID 17356139
- [Background] Miao K, Ni S, Zhou X, Xu N, Sun R, Zhuang C, Wang Y. Hidden blood loss and its influential factors after total hip arthroplasty. J Orthop Surg Res. 2015 Mar 18;10:36. doi: 10.1186/s13018-015-0185-9. PMID 25889223
- [Background] Levine BR, Haughom BD, Belkin MN, Goldstein ZH. Weighted versus uniform dose of tranexamic acid in patients undergoing primary, elective knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Sep;29(9 Suppl):186-8. doi: 10.1016/j.arth.2014.01.038. Epub 2014 May 27. PMID 24997651
- [Background] Zohar E, Ellis M, Ifrach N, Stern A, Sapir O, Fredman B. The postoperative blood-sparing efficacy of oral versus intravenous tranexamic acid after total knee replacement. Anesth Analg. 2004 Dec;99(6):1679-1683. doi: 10.1213/01.ANE.0000136770.75805.19. PMID 15562053
- [Background] Nilsson IM. Clinical pharmacology of aminocaproic and tranexamic acids. J Clin Pathol Suppl (R Coll Pathol). 1980;14:41-7. No abstract available. PMID 7000846
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD001886. doi: 10.1002/14651858.CD001886.pub3. PMID 21249650
- [Background] Poeran J, Rasul R, Suzuki S, Danninger T, Mazumdar M, Opperer M, Boettner F, Memtsoudis SG. Tranexamic acid use and postoperative outcomes in patients undergoing total hip or knee arthroplasty in the United States: retrospective analysis of effectiveness and safety. BMJ. 2014 Aug 12;349:g4829. doi: 10.1136/bmj.g4829. PMID 25116268
- [Background] Pleym H, Stenseth R, Wahba A, Bjella L, Karevold A, Dale O. Single-dose tranexamic acid reduces postoperative bleeding after coronary surgery in patients treated with aspirin until surgery. Anesth Analg. 2003 Apr;96(4):923-928. doi: 10.1213/01.ANE.0000054001.37346.03. PMID 12651635
- [Background] Weber CF, Gorlinger K, Byhahn C, Moritz A, Hanke AA, Zacharowski K, Meininger D. Tranexamic acid partially improves platelet function in patients treated with dual antiplatelet therapy. Eur J Anaesthesiol. 2011 Jan;28(1):57-62. doi: 10.1097/EJA.0b013e32834050ab. PMID 20962655
- [Background] He S, Johnsson H, Zabczyk M, Hultenby K, Cao H, Blomback M. A fibrinogen concentrate Haemocomplettan (Riastap) or a Factor XIII concentrate Fibrogammin combined with a mini dose of tranexamic acid can reverse the fibrin instability to fibrinolysis induced by thrombin- or FXa-inhibitor. Br J Haematol. 2013 Mar;160(6):806-16. doi: 10.1111/bjh.12189. Epub 2013 Jan 30. PMID 23360261
- [Background] Jansen AJ, Andreica S, Claeys M, D'Haese J, Camu F, Jochmans K. Use of tranexamic acid for an effective blood conservation strategy after total knee arthroplasty. Br J Anaesth. 1999 Oct;83(4):596-601. doi: 10.1093/bja/83.4.596. PMID 10673876
- [Background] Kim TK, Chang CB, Koh IJ. Practical issues for the use of tranexamic acid in total knee arthroplasty: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1849-58. doi: 10.1007/s00167-013-2487-y. Epub 2013 Mar 31. PMID 23542923
- [Background] Zhou XD, Tao LJ, Li J, Wu LD. Do we really need tranexamic acid in total hip arthroplasty? A meta-analysis of nineteen randomized controlled trials. Arch Orthop Trauma Surg. 2013 Jul;133(7):1017-27. doi: 10.1007/s00402-013-1761-2. Epub 2013 Apr 25. PMID 23615973
- [Background] Blanie A, Bellamy L, Rhayem Y, Flaujac C, Samama CM, Fontenay M, Rosencher N. Duration of postoperative fibrinolysis after total hip or knee replacement: a laboratory follow-up study. Thromb Res. 2013 Jan;131(1):e6-e11. doi: 10.1016/j.thromres.2012.11.006. Epub 2012 Nov 26. PMID 23195143
- [Background] Yamasaki S, Masuhara K, Fuji T. Tranexamic acid reduces blood loss after cementless total hip arthroplasty-prospective randomized study in 40 cases. Int Orthop. 2004 Apr;28(2):69-73. doi: 10.1007/s00264-003-0511-4. Epub 2003 Oct 10. PMID 15224162
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Background] Pilbrant A, Schannong M, Vessman J. Pharmacokinetics and bioavailability of tranexamic acid. Eur J Clin Pharmacol. 1981;20(1):65-72. doi: 10.1007/BF00554669. PMID 7308275
- [Background] Ekback G, Axelsson K, Ryttberg L, Edlund B, Kjellberg J, Weckstrom J, Carlsson O, Schott U. Tranexamic acid reduces blood loss in total hip replacement surgery. Anesth Analg. 2000 Nov;91(5):1124-30. doi: 10.1097/00000539-200011000-00014. PMID 11049894
- [Background] Soni A, Saini R, Gulati A, Paul R, Bhatty S, Rajoli SR. Comparison between intravenous and intra-articular regimens of tranexamic acid in reducing blood loss during total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1525-7. doi: 10.1016/j.arth.2014.03.039. Epub 2014 Apr 5. PMID 24814890
- [Background] Oremus K, Sostaric S, Trkulja V, Haspl M. Influence of tranexamic acid on postoperative autologous blood retransfusion in primary total hip and knee arthroplasty: a randomized controlled trial. Transfusion. 2014 Jan;54(1):31-41. doi: 10.1111/trf.12224. Epub 2013 Apr 25. PMID 23614539
- [Background] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Background] Gibon E, Courpied JP, Hamadouche M. Total joint replacement and blood loss: what is the best equation? Int Orthop. 2013 Apr;37(4):735-9. doi: 10.1007/s00264-013-1801-0. Epub 2013 Feb 6. PMID 23385607
- [Background] Napier RJ, Spence D, Diamond O, O'Brien S, Walsh T, Beverland DE. Modifiable factors delaying early discharge following primary joint arthroplasty. Eur J Orthop Surg Traumatol. 2013 Aug;23(6):665-9. doi: 10.1007/s00590-012-1053-5. Epub 2012 Jul 22. PMID 23412186
- [Background] Dawson J, Fitzpatrick R, Frost S, Gundle R, McLardy-Smith P, Murray D. Evidence for the validity of a patient-based instrument for assessment of outcome after revision hip replacement. J Bone Joint Surg Br. 2001 Nov;83(8):1125-9. doi: 10.1302/0301-620x.83b8.11643. PMID 11764424